CLINICAL TRIAL: NCT06541951
Title: Scale-up Implementation Approaches to Ending Pregnancy-related and -Associated Morbidity and Mortality (MIRACLE Center Project 3)
Brief Title: Scaling up Maternal Health Equity Best Practices
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jennifer E. Johnson, Chair, Charles Stewart Mott Department of Public Health, Michigan State University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00009307; U54HD113291 (NIH)
Record Dates: First submitted 2024-07-25; First posted 2024-08-07 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Maternal Mortality Disparities; Maternal Morbidity Disparities
Keywords: health inequities; maternal health; maternal mortality; implementation science; healthcare disparities; African Americans; Hispanic
MeSH Terms: conditions — Maternal Death

STUDY DESIGN:
Intervention Model Description: Cluster-randomized stepped wedge design
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Services as usual (Active Comparator): Services as usual before maternal health equity implementation efforts
  Interventions: Other: Services as usual
- Scale-up implementation approach (Experimental): An implementation approach for scaling up bundled equity-focused maternal health safety guidelines in community care settings county-wide, co-developed with partners.
  Interventions: Other: Scale-up implementation approach

INTERVENTIONS:
Other: Services as usual — During this phase of the stepped wedge design, agencies offering prenatal and postnatal care will follow their standard procedures
  Arms: Services as usual
Other: Scale-up implementation approach — An implementation approach for scaling up bundled equity-focused maternal health safety guidelines in community care settings county-wide, co-developed with partners. It may involve implementation approaches such as training, facilitation, learning collaboratives, coalitions, and other activities.
  Arms: Scale-up implementation approach

SUMMARY:
This study works with prenatal and postnatal care providers in 12 Michigan counties to scale up best practices for maternal health equity.

DETAILED DESCRIPTION:
The project recruits prenatal and postnatal care providers in 12 Michigan counties. his project will develop and test a scale-up focused implementation approach for addressing pregnancy-related and -associated morbidity and mortality (PRAMM) disparities. Previous efforts have shown that use of hospital- focused maternal safety bundles are an important part of successful efforts to reduce PRAMM. However, overall quality of obstetric care improved in these efforts without any effect on disparities. Thus, unlike previous efforts, the proposed project will implement quality improvement bundles that: (1) focus on PRAMM disparities; and (2) focus on community care (i.e., care provided outside the hospital in outpatient and other community settings) and coordination among care settings. Given that 83% of U.S. pregnancy-related and pregnancy-associated deaths occur during pregnancy or postpartum (rather than around the time of delivery), outpatient and community efforts are vital. Bundles (the evidence-based practices to be implemented) are developed by the national Alliance for Innovation on Maternal Health Community Care Initiative (AIM-CCI), and include "Community care for postpartum safety and wellness," and "Community care for maternal mental health," "Chronic conditions," and "Intimate partner violence" bundles. All bundles target PRAMM disparities. • Aim 1 of the proposed project will analyze bundle implementation experiences in 2 counties to develop a county-wide scale-up focused implementation approach for the bundles in partnership with stakeholders date to create and manualize a scale-up implementation intervention. • Aim 2 will evaluate the effectiveness and cost-effectiveness of the scale-up implementation intervention using a stepped wedge design in 12 Michigan counties with a total population of nearly 6 million people. PRAMM outcomes (individual level) will be extracted from a pre-existing statewide linked dataset. The sample for these analyses will include all Medicaid insured individuals in the 12 counties observed during pregnancy, at birth, and up to 1 year postpartum during the project period (~151,920 births, including ~49,110 births to African American and/or Hispanic mothers). Implementation outcomes (provider-level) include scale-up (penetration, reach, control for delivery, and intervention effectiveness at scale) and sustainment (maintenance of fidelity to core elements, health benefits, and capacity to deliver core elements over time). This project is innovative because it: (1) is the first controlled implementation trial to test approaches to implementing quality improvement bundles that: (a) specifically target PRAMM disparities; and (b) focus on community care; (2) advances the science of scale-up (it is the first study to test scale- up or sustainment implementation approaches to addressing maternal morbidity/mortality disparities); and (3) works to improve services across many (vs. a single) health systems. The project is significant because the field needs to reach pregnant people at scale, and scale-up is an understudied aspect of implementation science.

ELIGIBILITY:
Provider Inclusion Criteria:

-Be a provider or staff person at agencies offering prenatal and/or postnatal services in Wayne, Oakland, Ingham, Isabella, Macomb, Muskegon, Calhoun, Jackson, Saginaw, Kalamazoo, Barrien, or Washtenaw counties in Michigan.

Provider Exclusion Criteria:

* None

Patient outcomes are assessed through population-level Medicaid data, without direct recruitment.

Patient Inclusion criteria:

-All pregnant or postpartum (up to 12 months) people receiving Medicaid in Michigan

Patient Exclusion criteria:

-None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
African-American and Hispanic pregnancy-related and associated morbidity and mortality (PRAMM) | Continuous for 6 years
  A composite variable reflecting all pregnancy-related and associated morbidity and mortality conditions from pregnancy through 12 months postpartum, assessed using Medicaid claims data. The investigators will assess overall rates for African-American/Hispanic people and their rates relative to non-Hispanic white ones.

SECONDARY OUTCOMES:
Scale-up: Penetration | Assessed annually for 6 years
  Penetration (% providers/staff using recommended maternal health equity practices)
Scale-up: Reach | Assessed annually for 6 years
  Number of perinatal people receiving recommended practices
Scale-up: Control for delivery | Assessed annually for 6 years
  The degree to which control for delivery shifts to local actors and the practices are embedded in local delivery systems
Scale-up: Effectiveness | Assessed annually for 6 years
  Effectiveness is retained as the intervention is scaled: Operationalized using outcome 1 (PRAMM) analyses.
Sustainment: Fidelity | Annually for 6 years
  Fidelity to core elements at each time point as assessed through provider behavior assessed using a self-reported y/n responses to a checklist of activities
Sustainment: Health benefits | Annually for 6 years
  Health benefits continuing over time: Operationalized as the slope of PRAMM annually after the county moves into the "intervention phase of the stepped wedge design
Sustainment: Capacity | Annually for 6 years
  Capacity continues over time. Operationalized as the slope of capacity annually after the county moves into the "intervention" phase of the stepped wedge design
Cost of implementation approaches | Continuous over 6 years
  Cost via our grant accounting
Cost-effectiveness of implementation approaches | Continuous over 6 years
  The primary cost-effectiveness measure will be non-severe maternal morbidity, calculating intervention costs per point of score reduction. Secondary cost-effectiveness measures will be severe maternal morbidity and maternal mortality. Prevented severe maternal morbidity (SMM) will be also monetized using Medicaid claims data by calculating the difference between Medicaid delivery expenditures between women/birthing persons with SMM and without SMM using our own claims data and prior estimates. The value of a statistical life, currently around $10 million, will be used to monetize prevented maternal deaths.
Index (y/n) that is yes if there is any African-American and Hispanic severe maternal morbidity or pregnancy-associated mortality | Continuous for 6 years
  These will be assessed during pregnancy and through one-year postpartum using state Medicaid claims records and death records. The investigators will assess overall rates and rates relative to non-Hispanic white people.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E. Johnson, Ph.D., Principal Investigator — Michigan State University; Jaye Clement, MPH, MPP, Principal Investigator — Henry Ford Health; Amy Loree, PhD, Principal Investigator — Henry Ford Health
Locations (1):
- Michigan State University on behalf on 12 Michigan counties, Flint, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
The pre-existing statewide linked Medicaid dataset (individual level) is available from the Michigan Department of Health and Human Services, upon request, and with a new data use agreement to be initiated by the requesting individuals. Restrictions apply to the availability of these data, which were used under license for this study. De-identified implementation outcomes (provider level) data collected by the project will be available in appropriate national repositories and as well as by request from the PIs.

REFERENCES:
- [Derived] Johnson JE, Clement J, Sikorskii A, Loree A, Meulen MV, Roman L, Dearing JW, Bolder H, White JM, Sokol R, Meghea C. A cluster randomized stepped wedge implementation trial of scale-up approaches to ending pregnancy-related and -associated morbidity and mortality disparities in 12 Michigan counties: rationale and study protocol. Implement Sci Commun. 2025 Feb 20;6(1):19. doi: 10.1186/s43058-024-00677-7. PMID 39980059